CLINICAL TRIAL: NCT01077440
Title: Detection of Donor-Derived DNA in Semen Samples Among Recipients of Allogeneic Hematopoietic Stem-Cell Transplants
Brief Title: Presence of Donor-Derived DNA in Semen Samples From Cancer Survivors Who Underwent Donor Stem Cell Transplant
Status: Terminated | Type: Observational
Why Stopped: PI leaving institution
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Haydar Frangoul, Professor of Pediatrics, Vanderbilt University
Other Study IDs: CDR0000666593; P30CA068485 (NIH); VU-VICC-PED-0995
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Cancer Survivor; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Testicular Germ Cell Tumor
Keywords: cancer survivor; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; recurrent neuroblastoma; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III malignant testicular germ cell tumor; refractory multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Testicular Germ Cell Tumor; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Testicular Neoplasms | interventions — Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Your sample will only be used for research at Vanderbilt University and will not be sold. Health insurance companies and group health plans may not request your genetic information that comes from this research. As part of this study, we ask that the data from the semen analysis can be put into a databank at Vanderbilt and kept with data from other people in the study. Your data will be given a special code and will not identify you directly. We ask you to select yes or no to allow/disallow us to:
  * Use your semen sample for gene research.
  * Store/share your semen sample for future gene research in hematopoietic stem cell transplantation.
  * Store/share your semen sample for future gene research for other health problems (such as cancer, heart disease, etc).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men - age 18+
  Interventions: Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: flow cytometry; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA analysis — DNA analysis will be performed on samples collected.
Genetic: polymerase chain reaction — A polymerase chain reaction (PCR) assessment will be done on the samples collected.
Other: flow cytometry — Flow cytometry will be done on the samples collected.
Other: laboratory biomarker analysis — Laboratory biomarker analysis will be performed on the samples collected.

SUMMARY:
RATIONALE: Studying samples of semen from cancer survivors in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This phase I research study is looking at the presence of donor-derived DNA in semen samples form cancer survivors who underwent donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine semen samples from male survivors of allogeneic hematopoietic stem cell transplantation for the presence of donor-derived DNA.

OUTLINE: Semen samples are collected and assessed by flow cytometry and PCR. DNA samples are compared to previously analyzed DNA extracted from survivor and donor. Samples are also analyzed for sperm concentration, motility, morphology, and viability.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Disease in remission
* More than 365 days since prior allogeneic hematopoietic stem cell transplantation with history of full donor engraftment
* Stable complete donor chimerism

PATIENT CHARACTERISTICS:

* Able to consent and willing to provide a semen sample
* Survivors who present for long-term follow-up appointments in the adult and pediatric stem cell transplant clinic at Vanderbilt University Medical Center
* No known history of infertility or azospermia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No history of testicular irradiation ≥ 200 cGy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males over the age of 18 who have a history of allogeneic stem cell transplant >365 days ago with history of full donor engraftment, whose disease is in remission,
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Presence of donor-derived DNA in semen samples of male survivors of allogeneic hematopoietic stem cell transplantation | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Haydar A. Frangoul, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States